CLINICAL TRIAL: NCT04051164
Title: Effects of Progressive Muscle Relaxation Technique on Pulmonary Functions and Stress on Lower Limb Amputation
Brief Title: Progressive Muscle Relaxation Technique on Lower Limb Amputation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RiphahIU Khola Pervaiz
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Lower Limb Amputation Above Knee (Injury)
Keywords: Amputation; Progressive Muscle Relaxation Technique; Pulmonary Function; Stress
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Muscle Relaxation Technique (Experimental): Progressive muscle relaxation technique
  Interventions: Other: Progressive Muscle Relaxation Technique
- Conventional treatment (Active Comparator): Conventional Treatment: (Strengthening exercises of residual limb, Gait training, Deep Breathing exercise)
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Progressive Muscle Relaxation Technique — PMRT begins by assuming a comfortable position of lying down, sitting or leaning back.
  Patient is asked to take a breathe in and intentionally contract muscle and hold muscle and after that release all tension and focus on sensation of relaxation. Each muscle group is tensed for 5-7 seconds and relaxed for 20-30 seconds. PMRT is given twice a day for one week.
  Arms: Progressive Muscle Relaxation Technique
Other: Conventional treatment — Strengthening exercises of residual limb: After amputation strengthening exercises of residual limb is necessary to prevent shortening of muscles and tightening of joints, moreover it is necessary to make residual limb strong and flexible in order to use a prosthesis. This include Hip abduction, prone hip extension and Prone position. Gait training: This include standing exercises in the parallel bars with or without the prosthesis. Initial walking exercises in which the patient is taught to raise each knee alternately and to try to take weight on his limb as much as possible. Deep Breathing exercise: Deep breathing 10-15 repetitions twice a day.
  Arms: Conventional treatment

SUMMARY:
To determine the effects of progressive muscle relaxation technique on pulmonary functions in lower limb amputation patients. Randomized control Trail study design was chosen for this study, sampling technique Non probability convenient sampling then randomly allocated into groups by coin toss method. The subject in experimental group (n=20) were provided PMRT twice a day for one week and conventional treatment (n=20) was provided to control group. Modified perceived stress scale was used to find the effect of PMRT on stress, and pulmonary function was measured by digital spirometer..

DETAILED DESCRIPTION:
Normal functioning of cardiovascular system are controlled by autonomic nervous system. Stress causes autonomic imbalance which increases sympathetic activity. Loss of limb is potentially stressful change in one's life resulting in vast physical, occupational and psycho-social changes. Amputation is the removal of any part of body, when all other reconstructive strategies have failed. Lower limb amputation caused by diabetes annually costs between $30,000 to $60,000 and throughout life costs half a million dollar. It was estimated in 2012 that lower extremity wound and diabetes in U.S medicare program cost about $41 million dollar which is almost estimated as ~1.6 of all medicare health spending (1-4), however in U.K national health care spent almost an amount of £639 and 662 million on foot ulcers, which was approximately £1 in every £150 spent by the National Health Service.

Other studies done on cost of diabetic foot ulcer (DFU) in Belgium showed Us $10,572 and in Sweden total cost for healing was US$24,965/patient with no amputation while they were US $47,518 and US$42,858 with amputation with minor and major surgeries respectively. Amputation due to congenital deformity is les common and present in only 1% of total amputation done. Acquired amputations include Peripheral vascular disease, trauma, malignancy, metabolic and infection. 2 million people or even more in US are living with loss of limb, and accounts for 10 times more amputation in people with diabetes in comparison with those who don't have diabetes according to World health organization.

Musculoskeletal imbalances or pathologies often develop into secondary physical conditions or complications that may affect the mobility and quality of life of people with lower limb amputation. Using one or more prostheses causes people with amputation to alter the biomechanics of their movement. For example, people with lower-limb amputation often favor and stress their intact lower limb more during everyday activities.

This can lead to degenerative changes such as osteoarthritis of the knee and/or hip joints of the intact limb. Since people with amputation spend less time on their residual limb, osteopenia and subsequent osteoporosis often occur secondary to insufficient loading through the long bones of the lower limb. A proper prosthetic fit increases the probability of equal force distribution across the intact and prosthetic limbs during ambulation, thus decreasing the risk of osteoarthritis. People with limb loss commonly complain of back pain, which is linked to poor prosthetic fit and alignment, postural changes, leg-length discrepancy, amputation level, and general deconditioning. We review the literature on secondary complications among people with lower limb loss who are long-term prosthesis wearers.(outcomes of amputation) Secondary complications are of great importance in patients who have undergone traumatic amputation, main 2 systems that are effected are musculoskeletal and cardiovascular system. Mostly hospitalized patients acquire lying position which include spine, prone or right and left side lying position, change of position after every 2 hours is recommended to avoid contractures or bed sores, positioning is also required for good oxygen saturation and drainage of secretion, recumbency causes accumulation of secretions. Number of people having paraplegia and other disorders related to Central nervous system (CNS) are increasing due to metabolic disorder and increased blood pressure and most patients with CNS disorder are bed bound.

Estimation of pulmonary functions in various body postures they concluded that body position has a significant effect on spirometric measures like forced vital capacity (FVC), Forced expired volume in 1 second (FEV1) and FEV1%, generally. The standing position has highest lung volume and chair sitting to the second highest lung volumes. In recumbent position, factors causing impaired lung function include external compression of chest wall, compression of abdominal contents on diaphragm, compression of airway and blood vessels by heart.

Progressive muscle Relaxation Technique (PMRT) is one of the non pharmacological interventions to overcome these problems. It decreases stress through its effect on mental and physical conditions, mood, depression, and anxiety. Relaxation methods are very powerful tools for dealing with stress, depression and anxiety by giving the body/mind the chance to make its own healing.

Effect of of progressive muscle relaxation technique on Chronic Obstructive pulmonary Disease (COPD) patients and concluded that PMRT demonstrates an effective intervention approach for improving pulmonary function by reducing COPD-related fatigue and sleep quality.

Meta analysis on for collecting the evidence of effectiveness of relaxation techniques on pulmonary function of patients with COPD. They concluded that relaxation techniques improve oxygen saturation and heart rate therefore improving pulmonary function.

Randomized controlled trial on seventy two individuals with lung or gastrointestinal tumours to determine the effectiveness of relaxation techniques. It was concluded that progressive relaxation training is effective in improving fatigue and physical performance of cancer patients.

Prolong immobilization due to amputation badly effect pulmonary function, previously no study was done to know the effect of PMRT on pulmonary function. Effect of relaxation was seen in asthmatic children, asthma is a condition in which airway is narrowed, swell and produce extra mucus. For more than a period of 10 years it has been common place for physician and other dealing with asthmatic patients to ask them to relax at the onset of asthmatic attacks, there is no empirical data available but patient report and clinical experience suggested that relaxation can improve wheezing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Lower Limb amputation (up to level of trans femoral)immediate after surgery
* Single leg Amputated patients
* Both Genders.
* Amputation as a result of Diabetes Mellitus (DM) , trauma, burns and Electric Burn, Peripheral vascular disorders

Exclusion Criteria:

* Vitally unstable Patients.
* Patients with diagnosed respiratory disease.
* Any neurological Symptoms.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Forced vital Capacity (FVC) | 1 week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters
Forced Expiratory Volume in 1 second (FEV1) | 1 week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Peak Expiratory Flow (PEF) | 1 week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze peak expiratory flow PEF in Liter/second
Modified perceived stress scale | 2 week
  Perceived stress scale was developed in 1983, (36) and most commonly used to measure the degree to which situation in one's life are appraised as stressful. Modified perceived stress scale which consist of 10 items. Each item is rated on a 5-point scale ranging from never (0) to almost always (4).

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Tariq, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boulton AJ, Vileikyte L, Ragnarson-Tennvall G, Apelqvist J. The global burden of diabetic foot disease. Lancet. 2005 Nov 12;366(9498):1719-24. doi: 10.1016/S0140-6736(05)67698-2. PMID 16291066
- [Background] Margolis DJ, Jeffcoate W. Epidemiology of foot ulceration and amputation: can global variation be explained? Med Clin North Am. 2013 Sep;97(5):791-805. doi: 10.1016/j.mcna.2013.03.008. Epub 2013 Apr 25. PMID 23992892
- [Background] Feinglass J, Shively VP, Martin GJ, Huang ME, Soriano RH, Rodriguez HE, Pearce WH, Gordon EJ. How 'preventable' are lower extremity amputations? A qualitative study of patient perceptions of precipitating factors. Disabil Rehabil. 2012;34(25):2158-65. doi: 10.3109/09638288.2012.677936. Epub 2012 Apr 25. PMID 22533668
- [Background] Debigare R, Cote CH, Maltais F. Peripheral muscle wasting in chronic obstructive pulmonary disease. Clinical relevance and mechanisms. Am J Respir Crit Care Med. 2001 Nov 1;164(9):1712-7. doi: 10.1164/ajrccm.164.9.2104035. No abstract available. PMID 11719314
- [Background] Engelen MP, Schols AM, Does JD, Wouters EF. Skeletal muscle weakness is associated with wasting of extremity fat-free mass but not with airflow obstruction in patients with chronic obstructive pulmonary disease. Am J Clin Nutr. 2000 Mar;71(3):733-8. doi: 10.1093/ajcn/71.3.733. PMID 10702166
- [Background] Dehdari T, Heidarnia A, Ramezankhani A, Sadeghian S, Ghofranipour F. Effects of progressive muscular relaxation training on quality of life in anxious patients after coronary artery bypass graft surgery. Indian J Med Res. 2009 May;129(5):603-8. PMID 19675392
- [Background] Little BC, Hayworth J, Benson P, Hall F, Beard RW, Dewhurst J, Priest RG. Treatment of hypertension in pregnancy by relaxation and biofeedback. Lancet. 1984 Apr 21;1(8382):865-7. doi: 10.1016/s0140-6736(84)91337-0. PMID 6143184
- [Background] Akgun Sahin Z, Dayapoglu N. Effect of progressive relaxation exercises on fatigue and sleep quality in patients with chronic obstructive lung disease (COPD). Complement Ther Clin Pract. 2015 Nov;21(4):277-81. doi: 10.1016/j.ctcp.2015.10.002. Epub 2015 Oct 19. PMID 26573455
- [Background] Dimeo FC, Thomas F, Raabe-Menssen C, Propper F, Mathias M. Effect of aerobic exercise and relaxation training on fatigue and physical performance of cancer patients after surgery. A randomised controlled trial. Support Care Cancer. 2004 Nov;12(11):774-9. doi: 10.1007/s00520-004-0676-4. PMID 15338385